CLINICAL TRIAL: NCT03400085
Title: Pilot Study of a Mobile Health Intervention for Living Donor Follow-up
Brief Title: Pilot Study of an mHealth Intervention for Living Donor Follow-up
Acronym: mHealth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Texas Transplant Institute (Other); Vanderbilt University Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00162212; K01DK114388 (NIH)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Living Donors; Nephrectomy; Kidney
Keywords: mHealth; living donor kidney transplant; follow-up; health utilization

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized control trial with two arms. Participants in the intervention arm will use an mHealth application to complete their mandated living kidney donor follow-up at 6 months, 1 year, and 2 years, and participants in the control arm will receive the current standard of follow-up care and complete their required follow-up without the use of an mHealth application.
  Living Kidney Donors at the Vanderbilt University Medical Center are also being given the option to use the mKidney system, however, these study participants are not a part of the Pilot RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The control participants will be instructed to attend required follow-up as is standard of care, and will not receive the mHealth application.
- mHealth application (Experimental): Participants in the intervention arm will receive the mHealth application at their first post-donation clinic visit. Study personnel will assist participants assigned to the mHealth intervention arm with downloading the application and explain its functioning. Participants will then use the application to complete their required 6-month, 1-year, and 2-year follow-up.
  Interventions: Other: mHealth application

INTERVENTIONS:
Other: mHealth application — The intervention is an mHealth smartphone application designed for living kidney donors to complete their required 2-year follow-up. It allows the donor to input the answers to the clinical survey responses, as well as upload a picture of their lab values.
  Other Names: Application
  Arms: mHealth application

SUMMARY:
The investigators are interested in whether or not the use of a mobile health (mHealth) application increases the rate of follow-up compliance among living kidney donors. The investigators aim to test this by randomly assigning living kidney donors to the intervention (use of mHealth application to complete required living kidney donor follow-up at 6 months, 1 year, and 2 years) or control arm (standard of care) upon discharge from their initial donation hospitalization, and tracking follow-up compliance over time. The study population will be approximately 400 living kidney donors who undergo donor nephrectomy at Methodist Specialty and Transplant Hospital (200/year for 2 years).

The investigators will also recruit patients from the Vanderbilt University Medical Center into the study, however, these study participants are not a part of the Pilot Randomized Clinical Trial (RCT).

DETAILED DESCRIPTION:
Living kidney donation has been promoted as the 'best treatment option' for eligible patients with end-stage renal disease on the transplant waitlist by the American Society of Transplantation. In 2017, 5,264 living kidney donor (LKD) transplants were performed in the United States, representing over one-third of all kidney transplants performed nationally. While living donor nephrectomy is viewed as an overall safe procedure, the surgery does carry associated potential risks, including out-of-pocket costs, difficulty obtaining insurance, and long-term health complications. In 2013, the United Network for Organ Sharing (UNOS) passed new regulations requiring transplant hospitals to collect living kidney donor (LKD) follow-up data for a minimum of 2 years post-donation. Despite this national mandate, less than 50% of transplant hospitals were able to meet reporting thresholds for LKDs who donated in 2013. Documented challenges to collecting this data include cost, donor inconvenience, and data collection burden.

Therefore, novel methods are required to address incomplete donor follow-up. The investigators believe that mobile health (mHealth) systems, such as smartphone applications, would provide an effective, low-cost method of improving living donor follow-up rates. The investigators have built an mHealth system designed for reporting and collecting LKD follow-up data. The mHealth application was created based on previous studies conducted by the study team on the attitudes and perceptions of LKDs at a single transplant center on the use of mHealth for LKD follow-up, as well as after eliciting input from transplant thought leaders in the United States through semi-structured interviews. The aim of this study is to pilot test the mHealth system and compare the investigators' ability to achieve required follow-up at 6 months, 1 year, and 2 years against controls to help estimate potential effect sizes of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Have undergone live donor nephrectomy at Methodist Specialty and Transplant Hospital in San Antonio, Texas
* Have undergone live donor nephrectomy at Vanderbilt University Medical Center in Nashville, Tennessee

Exclusion Criteria:

* Participants will only be excluded if they do not consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month compliance to follow-up | 6 months
  Compliance with submitting questionnaires and laboratory values within 60 days of the six-month donation anniversary. Participants in the intervention arm will receive notifications when their follow-up is available to complete via the mHealth app, and subsequent notifications thereafter until either the donor completes both clinical and laboratory components of the required follow-up, or they are no longer compliant and within the 60-day window. Participants in the control arm will complete their follow-up as is current standard of care at Texas Transplant Institute.
1-year compliance to follow-up | 1 year
  Compliance with submitting questionnaires and laboratory values within 60 days of the 1-year donation anniversary. Participants in the intervention arm will receive notifications when their follow-up is available to complete via the mHealth app, and subsequent notifications thereafter until either the donor completes both clinical and laboratory components of the required follow-up, or they are no longer compliant and within the 60-day window. Participants in the control arm will complete their follow-up as is current standard of care at Texas Transplant Institute.
2-year compliance to follow-up | 2 years
  Compliance with submitting questionnaires and laboratory values within 60 days of the 2-year donation anniversary. Participants in the intervention arm will receive notifications when their follow-up is available to complete via the mHealth app, and subsequent notifications thereafter until either the donor completes both clinical and laboratory components of the required follow-up, or they are no longer compliant and within the 60-day window. Participants in the control arm will complete their follow-up as is current standard of care at Texas Transplant Institute.

SECONDARY OUTCOMES:
6-month center follow-up compliance | 6 months
  Overall center rate of compliance with follow-up with 80% of all donors within 60 days of the six-month donation anniversary.
1-year center follow-up compliance | 1 year
  Overall center rate of compliance with follow-up with 80% of all donors within 60 days of the 1-year donation anniversary.
2-year center follow-up compliance | 2 years
  Overall center rate of compliance with follow-up with 80% of all donors within 60 days of the 2-year donation anniversary.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Warren, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Methodist Specialty and Transplant Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaPointe Rudow D, Hays R, Baliga P, Cohen DJ, Cooper M, Danovitch GM, Dew MA, Gordon EJ, Mandelbrot DA, McGuire S, Milton J, Moore DR, Morgievich M, Schold JD, Segev DL, Serur D, Steiner RW, Tan JC, Waterman AD, Zavala EY, Rodrigue JR. Consensus conference on best practices in live kidney donation: recommendations to optimize education, access, and care. Am J Transplant. 2015 Apr;15(4):914-22. doi: 10.1111/ajt.13173. Epub 2015 Feb 3. PMID 25648884
- [Background] Organ Procurement and Transplantation Network. National Data 2017.
- [Background] Boyarsky BJ, Massie AB, Alejo JL, Van Arendonk KJ, Wildonger S, Garonzik-Wang JM, Montgomery RA, Deshpande NA, Muzaale AD, Segev DL. Experiences obtaining insurance after live kidney donation. Am J Transplant. 2014 Sep;14(9):2168-72. doi: 10.1111/ajt.12819. Epub 2014 Jul 16. PMID 25041695
- [Background] Rodrigue JR, Schold JD, Morrissey P, Whiting J, Vella J, Kayler LK, Katz D, Jones J, Kaplan B, Fleishman A, Pavlakis M, Mandelbrot DA; KDOC Study Group. Predonation Direct and Indirect Costs Incurred by Adults Who Donated a Kidney: Findings From the KDOC Study. Am J Transplant. 2015 Sep;15(9):2387-93. doi: 10.1111/ajt.13286. Epub 2015 May 5. PMID 25943721
- [Background] Segev DL, Muzaale AD, Caffo BS, Mehta SH, Singer AL, Taranto SE, McBride MA, Montgomery RA. Perioperative mortality and long-term survival following live kidney donation. JAMA. 2010 Mar 10;303(10):959-66. doi: 10.1001/jama.2010.237. PMID 20215610
- [Background] OPTN Policy 18 Living Donor Data Submission Requirements. 2016: 220.
- [Background] Henderson ML, Thomas AG, Shaffer A, Massie AB, Luo X, Holscher CM, Purnell TS, Lentine KL, Segev DL. The National Landscape of Living Kidney Donor Follow-Up in the United States. Am J Transplant. 2017 Dec;17(12):3131-3140. doi: 10.1111/ajt.14356. Epub 2017 Jun 30. PMID 28510355
- [Background] Ommen ES, LaPointe Rudow D, Medapalli RK, Schroppel B, Murphy B. When good intentions are not enough: obtaining follow-up data in living kidney donors. Am J Transplant. 2011 Dec;11(12):2575-81. doi: 10.1111/j.1600-6143.2011.03815.x. Epub 2011 Nov 4. PMID 22054024
- [Background] Mandelbrot DA, Pavlakis M. Living donor practices in the United States. Adv Chronic Kidney Dis. 2012 Jul;19(4):212-9. doi: 10.1053/j.ackd.2012.04.010. PMID 22732040
- [Background] Waterman AD, Dew MA, Davis CL, McCabe M, Wainright JL, Forland CL, Bolton L, Cooper M. Living-donor follow-up attitudes and practices in U.S. kidney and liver donor programs. Transplantation. 2013 Mar 27;95(6):883-8. doi: 10.1097/TP.0b013e31828279fd. PMID 23388736
- [Background] Mandelbrot DA, Pavlakis M, Karp SJ, Johnson SR, Hanto DW, Rodrigue JR. Practices and barriers in long-term living kidney donor follow-up: a survey of U.S. transplant centers. Transplantation. 2009 Oct 15;88(7):855-60. doi: 10.1097/TP.0b013e3181b6dfb9. PMID 19935453
- [Background] Fleming JN, Taber DJ, McElligott J, McGillicuddy JW, Treiber F. Mobile Health in Solid Organ Transplant: The Time Is Now. Am J Transplant. 2017 Sep;17(9):2263-2276. doi: 10.1111/ajt.14225. Epub 2017 Mar 17. PMID 28188681